CLINICAL TRIAL: NCT01010256
Title: The Expression of PTEN Protein and mRNA in Malignant Cells of Chronic Myelomonocytic Leukemia
Status: Terminated | Type: Observational
Why Stopped: PI moved institutions
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Other Study IDs: 111245
Record Dates: First submitted 2009-11-06; First posted 2009-11-09 (Estimated); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Chronic Myelomonocytic Leukemia
Keywords: To evaluate the phosphate and tension homolog deleted on chromosome ten (PTEN) protein level in leukemia cells from patients with CMML.; To identify the PTEN genetic defect in patients with deficient PTEN protein levels.; To evaluate the role of PTEN deregulation in CMML pathogenesis.
MeSH Terms: conditions — Leukemia, Myelomonocytic, Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Subjects diagnosed with CMML: Subjects ages 18 and older with a CMML diagnosis based on the WHO 2009 criteria, and who have signed an informed consent are eligible to participate in the study population of this clinical trial. A total of 12 patients will be consented.
- Control Group: The control group will consist of subjects ages 18 years or older who are healthy (i.e. no hematologic disorders) and have signed an informed consent. A total of 10 healthy control subjects will be consented.

SUMMARY:
The purpose of this study is to evaluate the level of a specific protein (PTEN) in the cancer cells of chronic myelomonocytic leukemia (CMML) patients. This protein might be involved in the transformation from normal blood cells to leukemia cells. The PTEN protein has not been investigated in CMML specifically but it has been discovered in closely related cancers. If this study demonstrates an abnormality in this protein, future testing will be designed to evaluate the genetic abnormality that resulted in lack of the normal presence of this protein. The goal is that the results of this study will help to develop new drugs and strategies to treat the future patients with CMML by understanding the abnormality of the disease at the cellular and molecular levels. The results of this study can also be utilized by future studies to develop individualized treatment to patients who have abnormal levels of this protein.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be at least 18 years or older.
* Subject must sign informed consent.
* For study population only, the subject must have a CMML diagnosis based on the WHO 2009 criteria.
* For control population only, the subject must be deemed healthy with no hematologic disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: During routine clinic visits, staff will present the option of participating in this clinical trial to eligible patients with a diagnosis of CMML. Also, healthy control patients will be asked to participate. The healthy control patients can be the subject's family members, friends, or volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2009-11-01 (Actual); Primary Completion 2019-10-03 (Actual); Study Completion 2019-10-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Emanuel, MD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States